CLINICAL TRIAL: NCT04623554
Title: Neo-train: Pre-operative Exercise During Neoadjuvant Chemotherapy in Patients With Breast Cancer - a Randomized Controlled Trial
Brief Title: Pre-operative Exercise During Neoadjuvant Chemotherapy in Patients With Breast Cancer
Acronym: Neo-train
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Danish Cancer Society (Other); University Hospital Southampton NHS Foundation Trust (Other); Region Zealand (Other); Naestved, Slagelse and Ringsted Hospitals (Unknown)
Responsible Party: Principal Investigator, Susanne Dalton, Professor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REG-074-2020
Record Dates: First submitted 2020-10-19; First posted 2020-11-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Prehabilitation; Pre-operative exercise; Breast cancer; Tumour regression; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with an intervention arm and a control arm
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not possible to blind the participants, care providers or investigators. However, the outcome assessors of the primary endpoint (MRI assessment) will not be informed of the patients' allocation. Further, the statistician and data manager are blinded as the group allocation will be coded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Prehabilitation program
  Interventions: Behavioral: Prehabilitation program
- Control arm (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Prehabilitation program — The prehabilitation program includes combined high-intensity interval training on a cycle ergometer and machine-based resistance exercise of large muscle groups supervised by a physiotherapist. Exercise sessions will take place in physiotherapy departments at local hospitals or in municipality rehabilitation centres 3 times a week during the neoadjuvant chemotherapy period and ending in the week before breast surgery (maximum estimated 29 weeks depending on number of chemotherapy cycles, dose delays and time of breast surgery). Participants will be screened for psychological distress four times and in case of moderate-severe distress be advised to visit the local Cancer Society Support Center where participants will be assessed and offered free services based on their psychosocial needs and available offers. Participation will be monitored.
  Arms: Intervention arm

SUMMARY:
The Neo-Train study is a randomized controlled trial investigating the effects of supervised pre-operative aerobic and resistance exercise in patients with breast cancer during neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The long neoadjuvant chemotherapy period in patients with breast cancer brings a time window of opportunity to investigate the potential of pre-operative exercise to increase treatment efficacy with improved tumour regression. A possible improvement in chemotherapy completion, lift in physical function, alleviated toxicities as well as changes in biological markers can also be investigated.

120 patients with newly diagnosed breast cancer who start neoadjuvant chemotherapy will be randomized to the intervention arm (n=60) and control arm (n=60).

Participants in the intervention arm will be prescribed a prehabilitation program consisting of thrice weekly combined supervised aerobic and resistance exercise during the neoadjuvant chemotherapy period. Participants will be screened for psychological distress four times and in case of moderate-severe distress be advised to visit the local Cancer Society Support Center where participants will be assessed and offered free services based on their psychosocial needs and available offers.

Participants in the control arm will receive usual care.

Outcomes will be measured at baseline (diagnosis), during neoadjuvant chemotherapy, during the week before breast surgery, at breast surgery and at 3 months follow up.

The participants will receive the recommended neoadjuvant chemotherapy regimens in Denmark - currently up to 24 weeks. With expected chemotherapy dose delays, the time of breast surgery is expected to be within 30 weeks from baseline. The treatment plans will be individually modified based on tumour response and expected side effects to treatment. A subgroup of participants may change neoadjuvant chemotherapy regimen and be referred to breast surgery early. In these participants, the last measurement during chemotherapy will be used, and the 3 months follow up measurement will still be scheduled at 3 months after breast surgery.

The study procedures will be pre-tested in a pilot study with 6 patients who will all receive the prehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with histologically verified breast cancer and scheduled for neoadjuvant chemotherapy
* Female gender
* Aged ≥ 18 years old
* Signed informed consent

Exclusion Criteria:

* Patients ineligible for or who have declined to receive neoadjuvant chemotherapy
* Contraindications to magnetic resonance imaging (MRI)
* Physical or cognitive disabilities preventing exercise or physical testing
* Inability to read and understand Danish
* Based on clinical judgement, the physician assesses that the patient is not suitable for inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2034-02-15 (Estimated)

PRIMARY OUTCOMES:
Tumour size | Sequential MRI scans follow the individual treatment plan in a period of up to 30 weeks from baseline (diagnostic MRI before start of neoadjuvant chemotherapy) to MRI performed by the end of the course of neoadjuvant chemotherapy before breast surgery.
  Change in the maximum diameter of the tumour visualized by magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Relative dose intensity of neoadjuvant chemotherapy | Baseline to time of breast surgery estimated up to 30 weeks
  Relative dose intensity in percentage defined as the ratio of received mg/m2 per week compared to planned mg/m2 per week according to standard guidelines.
Number of participants with neoadjuvant chemotherapy dose reductions | Baseline to time of breast surgery estimated up to 30 weeks
  Measured in percentage
Number of participants with neoadjuvant chemotherapy dose delays | Baseline to time of breast surgery estimated up to 30 weeks
  Measured in percentage
Number of participants with early discontinuation of neoadjuvant chemotherapy | Baseline to time of breast surgery estimated up to 30 weeks
  Measured in percentage
Number of hospital admissions during neoadjuvant chemotherapy | Baseline to time of breast surgery estimated up to 30 weeks
  Measured in percentage
Total length of hospital admissions during neoadjuvant chemotherapy | Baseline to time of breast surgery estimated up to 30 weeks
  Measured in days
Changes in total body mass | Baseline, during the week before breast surgery, 3 months after breast surgery
  Changes from baseline measured by bioelectrical impedance analysis.
Changes in lean body mass | Baseline, during the week before breast surgery, 3 months after breast surgery
  Changes from baseline measured by bioelectrical impedance analysis.
Changes in fat mass | Baseline, during the week before breast surgery, 3 months after breast surgery
  Changes from baseline measured by bioelectrical impedance analysis.
Changes in physical fitness | Baseline, week 13 during neoadjuvant chemotherapy, during the week before breast surgery, 3 months after breast surgery
  Changes in VO2 max estimated from maximum power output from baseline measured by a progressive cycle ergometer test (watt max test).
Changes in muscle strength | Baseline, week 13 during neoadjuvant chemotherapy, during the week before breast surgery, 3 months after breast surgery
  Changes in 1 repetition maximum strength from baseline measured on leg press and pull down.
Changes in physical function | Baseline, week 13 during neoadjuvant chemotherapy, during the week before breast surgery, 3 months after breast surgery
  Changes in hand grip strength from baseline measured by hand-held dynamometer in kilograms. Maximum kilograms obtained of 3 measurements on each hand.
Changes in level of physical activity | Baseline, during the week before breast surgery, 3 months after breast surgery
  Changes in activity data measured by a wearable objective measurement device.
Changes in health-related quality of life | Baseline, week 13 during neoadjuvant chemotherapy, during the week before breast surgery, 3 months after breast surgery
  Changes in self-reported health-related quality of life from baseline assessed on the Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B).
Changes in general anxiety | Baseline, week 13 during neoadjuvant chemotherapy, during the week before breast surgery, 3 months after breast surgery
  Changes in self-reported general anxiety from baseline assessed on the Generalised Anxiety Disorder 7-item (GAD-7).
Changes in depression | Baseline, week 13 during neoadjuvant chemotherapy, during the week before breast surgery, 3 months after breast surgery
  Changes in self-reported depression from baseline assessed on the Patient Health Questionnaire-9 (PHQ-9).
Changes in psychological distress | Baseline, week 13 during neoadjuvant chemotherapy, during the week before breast surgery, 3 months after breast surgery
  Changes in self-reported psychological distress from baseline assessed on the Distress Thermometer (DT).
Post-operative referral to and participation in municipal rehabilitation programs | Breast surgery to 3 months after breast surgery
  Frequency of participants referred to municipal rehabilitation, participation and types of activities attended identified from a self-reported questionnaire.
Tumour size | Sequential clinical examinations of the breast following the individual treatment plan in a period of up to 30 weeks from baseline to time of breast surgery
  Assessed by doctors' clinical examination of the breast.
Tumour size | At time of breast surgery estimated to take place within 30 weeks from baseline
  Measured by a pathologist from the tumour surgical specimen at breast surgery.
Pathological response grade | At time of breast surgery estimated to take place within 30 weeks from baseline
  Assessed by a pathologist from the tumour surgical specimen at breast surgery.
Tumour infiltrating lymphocyte population | Baseline (pre-chemotherapy) to time of breast surgery estimated up to 30 weeks
  Description of tumour infiltrating lymphocyte population (percentage of cells) evaluated by a pathologist from the tumour biopsy specimen taken before chemotherapy and tumour surgical specimen at breast surgery.
Tumour vascularity | Baseline (pre-chemotherapy) to time of breast surgery estimated up to 30 weeks
  Description of tumour vascularity density and structure evaluated by a pathologist from the tumour biopsy specimen taken before chemotherapy and tumour surgical specimen at breast surgery.
Liquid biopsies | Baseline, approximately week 7, 13 and 19, 3 months after breast surgery
  Changes in cell free DNA from blood samples. Furthermore, circulating tumour DNA will be investigated if possible.
Metabolic and inflammatory markers | Baseline, approximately week 13 and 19, 3 months after breast surgery
  Changes in glucose, hba1c, zinc, magnesium, phosphate and C reactive protein (CRP) levels from blood samples.
Cytokines | Baseline, approximately week 13 and 19, 3 months after breast surgery
  Changes in cytokines from blood samples before, during and after neoadjuvant chemotherapy.
Cell proliferation | Approximately between week 1-4 during neoadjuvant chemotherapy and within 6 weeks before breast surgery
  In vitro cell proliferation response with sera collected from blood samples before and after exercise.
Recurrence | Breast surgery to up to 10 years follow-up after breast surgery
  Incidence of breast cancer recurrence in percent
Survival | Breast surgery to up to 10 years follow-up after breast surgery
  Risk of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Dalton, Prof., Principal Investigator — Zealand University Hospital
Locations (1):
- Department of Clinical Oncology and Palliative Care, Zealand University Hospital, Næstved, Denmark

REFERENCES:
- [Background] Kjeldsted E, Ammitzboll G, Jorgensen LB, Lodin A, Bojesen RD, Ceballos SG, Rosthoj S, Laenkholm AV, Skou ST, Jack S, Gehl J, Dalton SO. Neo-train: study protocol and feasibility results for a two-arm randomized controlled trial investigating the effect of supervised exercise during neoadjuvant chemotherapy on tumour response in patients with breast cancer. BMC Cancer. 2023 Aug 19;23(1):777. doi: 10.1186/s12885-023-11284-5. PMID 37598196
- [Result] Kjeldsted E, Ammitzboll G, Laenkholm AV, Rasic D, Ceballos SG, Jorgensen LB, Skou ST, Bojesen RD, Lodin A, Tolver A, Rosthoj S, Jack S, Gehl J, Dalton SO. Effects of Supervised Exercise during Neoadjuvant Chemotherapy on Tumor Response in Patients with Breast Cancer (Neo-train): A Randomized Controlled Trial. Clin Cancer Res. 2025 Oct 15;31(20):4265-4277. doi: 10.1158/1078-0432.CCR-25-0416. PMID 40788186